CLINICAL TRIAL: NCT05147597
Title: Turkish Validity and Reliability of the Saint George Respiratory Questionnaire Idiopathic Pulmonary Fibrosis Version (SGRQ-I)
Brief Title: Turkish Validity and Reliability of SGRQ-I
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal investigator, Saglik Bilimleri Universitesi
Other Study IDs: TR_SGRQI
Record Dates: First submitted 2021-11-17; First posted 2021-12-07 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: IPF
Keywords: SGRQ; SGRQ-I; IPF; Quality of life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Cases diagnosed with Idiopathic pulmonary fibrosis (IPF) in the chest diseases outpatient clinic will be informed about the study, and the informed consent form will be signed by the specialist physician and demographic information will be obtained from the cases who accepted to be included in the study.
  The surveys will be contacted by the patient at 1-week intervals and answered by the patient by the responsible researcher and chest diseases physician.

SUMMARY:
The Saint George Respiratory Questionnaire (SGRQ) questionnaire is a frequently used questionnaire in the respiratory patient group, and the Turkish version of this questionnaire, which was created for use in idiopathic pulmonary fibrosis patients, is not available. There is no commonly used quality of life questionnaire in patients with idiopathic pulmonary fibrosis. The aim of the study is to translate and validate the SGRQ idiopathic pulmonary fibrosis version of questionnaire into Turkish.

DETAILED DESCRIPTION:
* The study is a cross-sectional, questionnaire validation study.
* It is planned to complete the study within 2 years after the sufficient sample size is reached and the evaluations are made. The study will be terminated when the sufficient number of patients is reached.
* The main thing in the application of special tools such as questionnaires is to prove the usability of the tool in the sample group to which it will be applied. The first step for this is the translation phase from the original language to the other language. At this stage, it is ideal for people who know the structure of the target language and the original language well, who have a good command of these languages and who are experienced in doing the translation. In our study, two people who are fluent in the original language will translate the questionnaire into the target language and two different people will translate the original language again.
* To the participants; Demographic Evaluation Form, Saint George's Respiratory Questionnaire (SGRQ), and SGRQ idiopathic pulmonary fibrosis version of Questionnaire (SGRQ-I) will be applied. The SGRQ-I questionnaire will be administered again one week after the first application date in order to determine the test-retest reliability.
* Scale reliability will be tested with Cronbach Alpha.For construct validity, confirmatory factor analysis will be applied and confirmatory factor analysis will be applied. For content validity, opinions of different experts will be taken for each item, and the status of items in the scale will be determined according to the results obtained by substituting it. In the logical validity process; Coverage of the components constituting the measured skill for each item will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Having a Diagnosis of Idiopathic Pulmonary Fibrosis
* To be literate in Turkish

Exclusion Criteria:

* Exacerbation or exacerbation in the last 6 weeks
* Presence of comorbidities affecting ambulation
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Turkish People
Study Population: Diagnosed with Idiopathic Pulmonary Fibrosis
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-01-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Saint George Respiratory Questionnaire - Idiopathic Pulmonary Fibrosis Version (SGRQ-I) | Change from baseline at 1 week.
  SGRQ-I consists of 34 self-complementing items. It was developed as an IPF-specific version of SGRQ. Different scales are used to score the SGRQ-I, resulting in an overall score and three domain scores: Effects, Activities, and Symptoms. Scores range from 0 to 100, with higher scores indicating more impaired health related quality of life.

SECONDARY OUTCOMES:
Saint George's Respiratory Questionnaire (SGRQ) | Change from baseline at 1 week.
  It is a 76-item questionnaire in which the total score and the three-component score are calculated. Components; symptoms (difficulty caused by symptoms such as cough, sputum, shortness of breath, and wheezing), activity (activity that causes or is limited by shortness of breath), and impact (social and psychological impact of the illness). Each item has its own weighted score. These weighted scores are not dependent on age, gender, disease duration and severity. It is not focused on a single language and culture. The evaluation feature of the questionnaire and its distinctiveness in different diseases and at different levels are high. Each of these scores ranges from 0 to 100. 0 indicates best health, 100 indicates worst health.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided